CLINICAL TRIAL: NCT04476641
Title: A Study of DC-CIK Immunotherapy in the Treatment of Solid Tumors
Acronym: DC-CIK
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jianchuan Xia, professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2016-036-02
Record Dates: First submitted 2020-07-10; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Liver Cancer; Kidney Cancer; Nasopharyngeal Cancer; Lung Cancer; Colorectal Cancer; Breast Cancer
MeSH Terms: conditions — Liver Neoplasms; Kidney Neoplasms; Nasopharyngeal Neoplasms; Lung Neoplasms; Colorectal Neoplasms; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DC-CIK (Experimental)
  Interventions: Other: CELL

INTERVENTIONS:
Other: CELL — inject the DC-CIK(dendritic cell activated and cytokine induced killer cell)

SUMMARY:
Main purpose of this study is through comparing with the external control, evaluation of autologous D - CIK cells immunotherapy to finish after conventional treatment of liver cancer, renal clear cell carcinoma and nasopharyngeal carcinoma, lung cancer, colon cancer, breast cancer patients with the clinical efficacy and safety of study population, including clinical liver, renal clear cell carcinoma and nasopharyngeal carcinoma, lung cancer, colon cancer, breast cancer after conventional treatment (surgery, chemotherapy and radiotherapy) patients.The primary outcome measures were overall survival and progression-free survival, while the secondary outcome measures were overall response rate and quality of life.

DETAILED DESCRIPTION:
This is a single center, single arm phase II clinical research, to evaluate the self D - CIK cells to treat liver cancer, renal clear cell carcinoma, nasopharyngeal carcinoma, lung cancer, colorectal cancer, breast cancer patient safety and efficacy of plan participants included 1372 cases of the subjects, experimental group 686 cases, control group 686 cases, control group adopts the liver, renal clear cell carcinoma, nasopharyngeal carcinoma, lung cancer, colorectal cancer, breast cancer patients after conventional treatment (surgery, chemotherapy and radiotherapy) did not receive D - CIK cell therapy of external control

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients diagnosed with liver cancer, renal clear cell carcinoma, nasopharyngeal carcinoma, lung cancer, colorectal cancer, breast cancer and nasopharyngeal carcinoma by imaging examination, tissue and/or cytology, and patients after conventional treatment (surgery, chemotherapy and radiotherapy); (2) No history of other tumors (except surgically cured skin squamous cell carcinoma).

  (3) Male or female, aged over 18 and under 75 (including 18 and 75 years old). (4) Physical condition: ECOG score 0 or 1. (5) Expected survival time ≥ 6 months, and follow-up was available. (6) Within 7 days before the start of treatment, the results of blood routine, liver and kidney function, and hemagglutination laboratory examination meet the following standards:White blood cell (WBC) ≥ 3.5×109/L, platelet (PLT) ≥ 80×109/L, Neutropene (ANC) ≥ 1.5×109/L, hemoglobin (HGB) ≥ 90g/L, aspartic acid transaminase (AST) < 2.5× normal upper limit (ULN) (liver metastasis < 5×ULN), alanine transaminase (ALT) < 2.5×ULN (liver metastasis < 5×ULN), total bilirubin (TIBC) < 1.5×ULN,Serum creatinine (CR) < 1.0×ULN, prothrombin time, partial thrombin time, plasma fibrinogen, thrombin time were within the normal range.

  (7) Female subjects must use effective contraceptives (such as prescription oral contraceptives, injectable contraceptives, iUDS, double blocking, contraceptive patch, male partner sterilization, etc.) throughout the study period;Serum or urine pregnancy test results must be negative during screening and throughout the study period.

  (8) Male subjects should take effective contraceptive measures within 1 month after receiving treatment and completing chemotherapy.

  (9) Be willing to comply with the prohibitions and restrictions stipulated in the research plan.

  (10) The subjects have signed an informed consent, stating that they understand the purpose, procedure and content of the study and are willing to participate in the study.

Exclusion Criteria:

* (1) Patients with clinical symptoms of brain metastasis (except after radiotherapy).

  (2) There is an active viral or bacterial infection that cannot be controlled with appropriate anti-infective therapy.

  (3) Known to be serologically positive for HIV, syphilis, active HBV or HCV infection.

  (4) Having a mental illness or other medical condition, such as uncontrollable heart or lung disease, diabetes, etc., and failing to comply with the requirements of research treatment and monitoring.

  (5) Those who are known to be allergic to any component in cultured D-CIK cells.

  (6) Active rheumatic diseases. (7) Organ transplanters. (8) Poor compliance. (9) Women during pregnancy. (10) Lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 686 (Estimated)
Dates: Start 2016-05-06 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
OS and PFS | The enrollment period was 3 years and the follow-up period was 5 years
  Overall survival and progression-free survival

SECONDARY OUTCOMES:
ORR, CR+PR | The enrollment period was 3 years and the follow-up period was 5 years
  Overall response rate and quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Jianchuan Xia, Study Director — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No